CLINICAL TRIAL: NCT01463033
Title: Pilot: Levetiracetam to Prevent Post-Traumatic Epilepsy
Brief Title: Levetiracetam to Prevent Post-Traumatic Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pavel Klein (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor-Investigator, Pavel Klein, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NS45656
Record Dates: First submitted 2011-10-12; First posted 2011-11-01 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy; Post-traumatic Epilepsy
Keywords: Post-Traumatic epilepsy; Traumatic brain injury; Epilepsy prevention; Levetiracetam
MeSH Terms: conditions — Epilepsy; Epilepsy, Post-Traumatic; Brain Injuries, Traumatic | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levetiracetam (Active Comparator): 66 subjects with acute head injury with a high risk for developing post-traumatic epilepsy will receive levetiracetam 55 mg/kg/day in a b.i.d. schedule. Treatment will commence within 8 hours of the acute head injury and will last for 30 days. In addition, subjects will receive phenytoin for 1 week following head injury as standard clinical care.
  Interventions: Drug: Levetiracetam
- No Intervention Control (No Intervention): 60 subjects with acute head injury with a high risk for developing post-traumatic epilepsy enrolled 8-24 hours after injury will not receive levetiracetam. Subjects will receive phenytoin for 1 week following head injury as standard clinical care.

INTERVENTIONS:
Drug: Levetiracetam — 55 mg/kg/day given in 2 divided doses 12 hours apart
  Other Names: Keppra (brand name)
  Arms: Levetiracetam

SUMMARY:
Head injury is the cause of approximately 5% of all epilepsy in the US. Past attempts at preventing epilepsy by treatment with older antiepileptic drugs have been unsuccessful. Levetiracetam is a novel AED with potent antiepileptogenic properties in animal models of epilepsy. It has a favorable side effect and pharmacokinetic profile. It is therefore a strong candidate for a clinical trial of epilepsy prevention following traumatic brain injury (TBI). However, there has been no experience in administering levetiracetam rapidly to individuals with acute TBI. The investigators propose to initiate the evaluation of levetiracetam in prevention of post-traumatic epilepsy by determining the safety, tolerability, pharmacokinetics and feasibility of acute and chronic administration of levetiracetam to individuals with head injury with a high risk for developing post-traumatic epilepsy. Further, the investigators will follow subjects for 2 years after injury in order to obtain pilot data about effect of levetiracetam on PTE. This pilot study is the first step in evaluation of levetiracetam in prevention of post-traumatic epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Acute head injury associated with one of the following:

Intracranial hemorrhage, including epidural, subdural and intracerebral hemorrhage or with cerebral contusion(s) of any size; Penetrating (foreign body) head injury; Skull fracture and dural tear; Seizure within 8 hours of head injury

* Onset of head injury within 8-hours of proposed treatment initiation.
* Glasgow Coma Scale 6-15.

Exclusion Criteria:

* Clinical contraindications:

  * Previous epilepsy or status epilepticus.
  * Any systemic illness or unstable medical condition that might pose additional risk, including: renal insufficiency, other unstable metabolic or endocrine disturbances, and active systemic cancer.
  * Psychosis within six months of enrollment as determined by history of hospitalization for psychosis or medications for psychosis.
  * Moderate to severe mental retardation (IQ< 55 or>2 school grade levels below the expected for age [expected age = grade level +5]).
* Clinical/Laboratory Indicators:

  * Serum creatinine > 1.5 on the day of treatment initiation for adults.
  * Serum creatinine ≥1.5 for subjects ≥17 years old, ≥1.0 for subjects 13-17 years old and ≥0.7 for subjects 6-12 years old.
  * Pregnancy
  * Use of any CNS-active investigational drugs within 3 months of enrollment.
  * Use of Antiepileptic Drugs (AEDs) within two months of enrollment, for any indication.
  * Allergy/sensitivity to study drugs or their formulations:
  * Active drug or alcohol dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements:
  * Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, M.D., Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - MedStar Research Institute, Washington D.C., District of Columbia

REFERENCES:
- [Result] Pearl PL, McCarter R, McGavin CL, Yu Y, Sandoval F, Trzcinski S, Atabaki SM, Tsuchida T, van den Anker J, He J, Klein P. Results of phase II levetiracetam trial following acute head injury in children at risk for posttraumatic epilepsy. Epilepsia. 2013 Sep;54(9):e135-7. doi: 10.1111/epi.12326. Epub 2013 Jul 22. PMID 23876024
- [Result] Klein P, Herr D, Pearl PL, Natale J, Levine Z, Nogay C, Sandoval F, Trzcinsky S, Atabaki SM, Tsuchida T, van den Anker J, Soldin SJ, He J, McCarter R. Results of phase II pharmacokinetic study of levetiracetam for prevention of post-traumatic epilepsy. Epilepsy Behav. 2012 Aug;24(4):457-61. doi: 10.1016/j.yebeh.2012.05.011. Epub 2012 Jul 7. PMID 22771222
- [Result] Klein P, Herr D, Pearl PL, Natale J, Levine Z, Nogay C, Sandoval F, Trzcinski S, Atabaki SM, Tsuchida T, van den Anker J, Soldin SJ, He J, McCarter R. Results of phase 2 safety and feasibility study of treatment with levetiracetam for prevention of posttraumatic epilepsy. Arch Neurol. 2012 Oct;69(10):1290-5. doi: 10.1001/archneurol.2012.445. PMID 22777131

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational: 60 subjects with acute head injury with a high risk for developing post-traumatic epilepsy enrolled 8-24 hours after injury will not receive levetiracetam. Subjects will receive phenytoin for 1 week following head injury as standard clinical care.
Period: Overall Study
Arm/Group | Levetiracetam | Observational
Started | 66 | 60
Completed | 59 (3 deaths, 4 lost to follow up) | 54 (2 deaths, 4 lost to follow up)
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 4 | 4
Not completed — Death | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | Observational | Total
Number analyzed (Participants) | 66 | 60 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 41 | 33 | 74
  >=65 years | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Post-Traumatic Epilepsy
Description: occurrence of PTE (Post-Traumatic Epilepsy)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Levetiracetam | Observational
Number analyzed (Participants) | 66 | 60
participants | 6 | 8

2. Secondary Outcome: Adverse Events
Description: The 66 subjects with acute head injury with a high risk for developing post-traumatic epilepsy that received levetiracetam 55 mg/kg/day in a b.i.d. were monitored for adverse events through the 30 day treatment period.
Time Frame: 30 day treatment period
Population: The 66 subjects with acute head injury with a high risk for developing post-traumatic epilepsy that received levetiracetam 55 mg/kg/day in a b.i.d. were monitored for adverse events through the 30 day treatment period. Symptoms reported to be moderate or severe are listed. Adverse events were not monitored for the Observational group.
Measure: Number; unit: Events
Groups:
- Participants: The 66 subjects with acute head injury with a high risk for developing post-traumatic epilepsy that received levetiracetam 55 mg/kg/day in a b.i.d. schedule were monitored for adverse events through the 30 day treatment period.
Arm/Group | Participants
Number analyzed (Participants) | 66
Events
  Headache | 28
  Fatigue | 28
  Drowsiness | 20
  Memory Impairment | 9
  Amnesia | 8
  Pain | 15
  Irritability | 10
  Dizziness | 10
  Anorexia | 6
  Emotional lability | 7
  Insomnia | 5
  Cognitive changes | 7
  Ataxia | 6
  Depression | 7
  Hostility | 3
  Vertigo | 1
  Nausea | 2
  Cough | 2
  Nervousness | 5
  Paraesthesia | 3
  Weight gain | 1
  Hallucinations | 5
  Other | 2
  Diplopia | 3
  Suicidality | 3
  Psychosis | 3

ADVERSE EVENTS:
Time Frame: 30 day treatment period
Description: The 66 subjects with acute head injury with a high risk for developing post-traumatic epilepsy that received levetiracetam 55 mg/kg/day in a b.i.d. were monitored for adverse events through the 30 day treatment period. Adverse events were not monitored for the Observational group.
Groups:
- Levetiracetam: The 66 subjects with acute head injury with a high risk for developing post-traumatic epilepsy that received levetiracetam 55 mg/kg/day in a b.i.d. were monitored for adverse events through the 30 day treatment period. Adverse events were not monitored for the Observational group.
- Observational: Adverse events were not monitored for the Observational group
Arm/Group | Levetiracetam | Observational
Serious Adverse Events (participants affected / at risk) | 18/66 | 0/0
Other Adverse Events (participants affected / at risk) | 66/66 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=66) | Observational (N=0)
Depression (Psychiatric disorders) | 7 (7) | 0 (0)
Halluscinations (Psychiatric disorders) | 5 (5) | 0 (0)
Suicidality (Psychiatric disorders) | 3 (3) | 0 (0)
Psychosis (Psychiatric disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=66) | Observational (N=0)
Headache (Nervous system disorders) | 28 (28) | 0 (0)
Fatigue (General disorders) | 28 (28) | 0 (0)
Drowsiness (Nervous system disorders) | 20 (20) | 0 (0)
Memory Impairment (Nervous system disorders) | 9 (9) | 0 (0)
Amnesia (Nervous system disorders) | 8 (8) | 0 (0)
Pain (General disorders) | 15 (15) | 0 (0)
Irritability (General disorders) | 10 (10) | 0 (0)
Dizziness (Nervous system disorders) | 10 (10) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 7 (7) | 0 (0)
Ataxia (Nervous system disorders) | 6 (6) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Weight Gain (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No